CLINICAL TRIAL: NCT06509308
Title: The Role of Expectations in Chronic Obstructive Pulmonary Disease (COPD) - Development and Validation of a New Tool
Brief Title: Illness Expectations in COPD
Acronym: ASPECTO-BPCO
Status: Recruiting | Type: Observational
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Eleonora Volpato, Clinical Professor, Fondazione Don Carlo Gnocchi Onlus
Other Study IDs: FDG 88-18
Record Dates: First submitted 2024-04-06; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; Clinical Psychology; Rehabilitation Psychology; Chronic Illness
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Psychological Questionnaires — Patients will be asked to complete a series of questionnaires regarding disease expectations, cognitions, and representations of their health status. Additionally, sociodemographic data and clinical variables will be collected from medical records.

SUMMARY:
This study investigates the impact of expectations on individuals with Chronic Obstructive Pulmonary Disease (COPD) and aims to develop and validate a novel tool to assess these expectations. By understanding the role of expectations, healthcare providers can better tailor interventions and support for COPD patients, ultimately improving their quality of life and treatment outcomes.

DETAILED DESCRIPTION:
This research, carried out at the specialized cardiorespiratory rehabilitation unit of the Don Gnocchi Foundation in Milan, delves into the influence of expectations on individuals living with Chronic Obstructive Pulmonary Disease (COPD). The primary objective is to craft and validate a fresh assessment tool to gauge these expectations. Moreover, the questionnaire is reintroduced to patients after a month, during which additional data, as detailed in the corresponding section, are gathered.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD confirmed by spirometry
* Adults
* Italian speakers
* Ability to complete the required tests
* Informed consent from the patient to participate in the study

Exclusion Criteria:

* Non-Italian speakers
* Psychiatric comorbidities
* Cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients involved in the study are from the cardio-respiratory rehabilitation department of the Don Gnocchi Foundation in Milan. They have a confirmed diagnosis of COPD, with the severity level specified according to guidelines (thus, patients with mild, moderate, severe, or very severe COPD are included). Both male and female patients of any age are admitted, provided they are adults. Patients may have other respiratory and non-respiratory conditions, as long as they are documented. Individuals who do not understand the Italian language or who exhibit psychiatric comorbidities or cognitive impairment cannot be included.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Chronic Obstructive Pulmonary Disease Expectations Questionnaire | From October 2023 to January 2025
  A questionnaire composed of 27 items, designed by us, asking the patient to assess their disease expectations for the next 3 months. Each item is rated on a 7-point Likert scale, allowing for a nuanced evaluation of the patient's perceptions and expectations. Scores range from 27 to 189. A higher score indicates a worse illness perception.
  A questionnaire composed of 27 items, designed by us, asking the patient to assess their disease expectations for the next 3 months. Each item is rated on a 7-point Likert scale, allowing for a nuanced evaluation of the patient's perceptions and expectations. Scores range from 27 to 189. A higher score indicates a worse illness perception.

SECONDARY OUTCOMES:
Socio-demographic variables | From October 2023 to January 2025
  Gender, age, smoking status, and number of cigarettes smoked per day. Additionally, factors such as family history of respiratory diseases, alcohol use (frequency), physical activity (frequency and type), level of education, marital status, onset of initial symptoms, and date of diagnosis will be considered.
Body Mass Index | From October 2023 to January 2025
  kg/m^2
Medical data | From October 2023 to January 2025
  parameters from respiratory function tests (particularly Forced Vital Capacity (FVC) and Diffusing Capacity of the Lungs for Carbon Monoxide (DLCO), arterial blood gas analysis) will be recorded. These data will be extracted from the latest available medical report and therefore from the last pulmonary visit conducted as part of routine clinical practice (please note that medical visits paid for by this project are not included).
Brief Illness Perception Questionnaire | From October 2023 to January 2025
  The BIPQ is self-report questionnaire consisting of 8 items, rated on a 10-point Likert scale, investigates perceptions of illness (representations of cause, consequence, identity, control, duration), and requires the patient to nominate 3 factors they believe triggered the illness. The total score is calculated by summing the scores of all items, with a possible range of 0-80. Higher scores indicate worse illness perception. <42 indicating low experienced threat, 42-49 indicating moderate experienced threat, and ≥50 indicating high experienced threat in patients with a recently acquired spinal cord injury.
Illness Cognition Questionnaire | From October 2023 to January 2025
  The ICG is a 18-item questionnaire that contains three 6-item scales related to the factors helplessness, acceptance and perceived benefits, each with a scoring range of 6-24 Helplessness (items 1, 5, 7, 9, 12, 15), Acceptance (items 2, 3, 10, 13, 14, 17), and Perceived Benefits (items 4, 6, 8, 11, 16, 18).
Chronic Obstructive Pulmonary Disease Assessment TEST | From October 2023 to January 2025
  The CAT is a self-report questionnaire consisting of 8 items, rated on a 6-point Likert scale, where patients are asked to rate COPD impact on their quality of life. Range of CAT scores from 0-40. Higher scores denote a more severe impact of COPD on a patient's life. Scores <10 have a low impact, 10-20 medium, 21-30 high and >30 very high impact
Pharmacological Therapy | From October 2023 to January 2025
  A list of the medications taken by the patient.
Comorbidities | From October 2023 to January 2025
  A list of the major illness suffered from the patient.
Exacerbations and hospitalizations | From October 2023 to January 2025
  frequency of exacerbations and hospitalizations over the past year

CONTACTS AND LOCATIONS:
Locations (1):
- Don Gnocchi Foundation, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pagnini F. The potential role of illness expectations in the progression of medical diseases. BMC Psychol. 2019 Nov 8;7(1):70. doi: 10.1186/s40359-019-0346-4. PMID 31703607
- [Result] Rennard SI. COPD: overview of definitions, epidemiology, and factors influencing its development. Chest. 1998 Apr;113(4 Suppl):235S-241S. doi: 10.1378/chest.113.4_supplement.235s. PMID 9552012
- [Result] Kaptein AA, Scharloo M, Fischer MJ, Snoei L, Cameron LD, Sont JK, Rabe KF, Weinman J. Illness perceptions and COPD: an emerging field for COPD patient management. J Asthma. 2008 Oct;45(8):625-9. doi: 10.1080/02770900802127048. PMID 18951252
- [Result] Evers AW, Kraaimaat FW, van Lankveld W, Jongen PJ, Jacobs JW, Bijlsma JW. Beyond unfavorable thinking: the illness cognition questionnaire for chronic diseases. J Consult Clin Psychol. 2001 Dec;69(6):1026-36. PMID 11777106
- [Result] Broadbent E, Petrie KJ, Main J, Weinman J. The brief illness perception questionnaire. J Psychosom Res. 2006 Jun;60(6):631-7. doi: 10.1016/j.jpsychores.2005.10.020. PMID 16731240